CLINICAL TRIAL: NCT00582634
Title: Phase II Study of Adjuvant Cisplatin and Docetaxel in Non-small Cell Lung Cancer
Brief Title: Adjuvant Cisplatin and Docetaxel in Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2004-0248; CO04503 (Other: University of Wisconsin Carbone Cancer Center); H-2004-0248 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH/MEDICINE (Other: UW Madison)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2015-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: non small cell lung cancer; adjuvant; cisplatin; docetaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel followed by cisplatin (Experimental): Docetaxel (75mg/m2) given IV followed by cisplatin (75mg/m2) given IV on day 1 of a 21 day cycle. Both drugs will be administered intravenously over 1 hour each for 4 cycles.
  Interventions: Drug: docetaxel and cisplatin

INTERVENTIONS:
Drug: docetaxel and cisplatin — Docetaxel (75mg/m2) followed by cisplatin (75mg/m2) on day 1 of a 21 day cycle. Both drugs will be administered intravenously over 1 hour each for4 cycles.
  Other Names: Taxotere

SUMMARY:
* To determine if docetaxel and cisplatin can be administered in a dose intense manner in the adjuvant setting in resected non-small cell lung cancer
* To evaluate the time to progression and overall survival
* To evaluate toxicities of this chemotherapy combination in the adjuvant setting
* To correlate XPD and ERCC1 polymorphisms with time to progression and toxicities in patients treated with this regimen

ELIGIBILITY:
Inclusion Criteria:

* Stage IB to IIIA non-small cell lung cancer completely resected within 4 to 8 weeks of initiating treatment on study
* Performance Status ECOG 0 or 1
* Peripheral neuropathy: < grade 1
* Adequate blood cell counts
* Adequate liver and hepatic function
* Women of childbearing potential must have a negative pregnancy test.
* Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter

Exclusion Criteria:

* Patients with a history of severe hypersensitivity reaction to Docetaxel® or other drugs formulated with polysorbate 80.
* Women who are breast-feeding.
* Coexistent second malignancy or history of prior malignancy within previous 5 years (excluding basal or squamous cell carcinoma of the skin that has been treated curatively)
* Uncontrolled cardiac disease or uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2004-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Time to progression | 36 months
Overall survival | 36 months
Incidence of adverse events | Baseline to 36 months

SECONDARY OUTCOMES:
Correlate XPD and ERCC1 polymorphisms with time to progression and toxicities | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Traynor, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu